CLINICAL TRIAL: NCT02417077
Title: Perception of Facial Expression in Subjects With and Without Crow's Feet Lines
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: GMA-BTXC-14-001
Record Dates: First submitted 2015-04-10; First posted 2015-04-15 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Photographic Review: Photographic review of subjects who received treatment with onabotulinumtoxinA for crow's feet lines.
  Interventions: Other: Photographic Review

INTERVENTIONS:
Other: Photographic Review — Photographic review of subjects who received treatment with onabotulinumtoxinA for crow's feet lines.
  Other Names: BOTOX® Cosmetic

SUMMARY:
This study will examine the perception of facial expressions among individuals with and without crow's feet lines.

ELIGIBILITY:
Inclusion Criteria:

* English fluency

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 393 (Actual)
Dates: Start 2015-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Independant Observers' Perception of Expressed Emotions on a 7-Point Scale | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Saratoga Springs, New York, United States